CLINICAL TRIAL: NCT00184730
Title: Investigation of the Efficacy and Safety of hGH in Long Term (More Than 48 Weeks) in GHDA.
Brief Title: Long-term Trial on Growth Hormone Deficiency in Adults (GHDA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHLIQUID-1650; JapicCTI-050134 (Registry Identifier: japic)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Japan. This protocol describes an extension trial to supply hGH to subjects who wish continuous treatment after the long-term Phase 3 trial (GHLiquid-1519) until hGH products have been approved for GHDA in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed GHLiquid-1519.
* If the subject has a history of treatment for a tumor of pituitary or peripheral site, two years or more have to be passed since completion of surgery, radiotherapy or other treatment, and recurrence of the underlying disease to be excluded.
* Appropriate replacement therapy has been administered for more than 24 weeks for the treatment of other pituitary hormone deficiencies.

Exclusion Criteria:

* Subject with a history of acromegaly.
* Subject with diabetes mellitus.
* Subject suffering from malignancy.
* Several medical conditions

Ages: 19 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Lipid-related laboratory tests parameters (total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglyceride) | at the end of treatment
GH-related laboratory parameters (IGF-I, IGF-I SDS, IGFBP-3, IGFBP-3 SDS and IGF-I / IGFBP-3 molar ratio) | at the end of treatment

SECONDARY OUTCOMES:
Adverse events
FPG, insulin, and HbA1C
Clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com